CLINICAL TRIAL: NCT04425473
Title: Effect of Esketamine on Perioperative Depressive Symptoms in Patients Undergoing Major Surgery
Brief Title: Esketamine and Perioperative Depressive Symptoms
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Ruquan Han, Professor, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Z191100006619067
Record Dates: First submitted 2020-06-08; First posted 2020-06-11 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Depressive Symptoms; Esketamine; Perioperative Complication; Major Surgery
MeSH Terms: conditions — Depression | interventions — Esketamine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Esketamine (Experimental)
  Interventions: Drug: Esketamine
- Placebo (Placebo Comparator)
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Esketamine — Esketamine will be administrated intravenously when suturing incision, with total dose of 0.2mg/kg and continuous infusion for 40 minutes.
  Arms: Esketamine
Drug: Normal saline — Equivalent amount of normal saline will be administrated intravenously suturing incision.
  Arms: Placebo

SUMMARY:
Perioperative depressive symptoms (PDS) are common in population undergoing surgery, and this would be sharpened especially for complicated, high-risk major surgery. However, None of treatments could resolve this clinical problem during limited perioperative period. The remarkable effects of ketamine on treatment resistant depression have been verified by several clinical trials and the enantiomer S-ketamine (esketamine) showed similar antidepressant efficacy with better safety in recent studies. The efficacy and safety of esketamine administrated intra-operatively for PDS will be verified in this study. Other secondary outcomes such as anxiety, postoperative pain and psychiatric symptoms will also be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Patient undergoing elective major surgery
* Ages between 18 and 65 years old
* Moderate to severe depressive symptoms ( the Patient Health Questionnaire-9 scores equal to or more than 10 and Montgomery-Åsberg Depression Rating Scale scores equal to or more than 22 )
* Signed informed consent

Exclusion Criteria:

* had aphasia or any conditions that prevented mental health assessments,
* had a history of psychotic or bipolar disorder,
* had a comorbidity that affected hormone levels,
* required prolonged postoperative mechanical ventilation,
* had received treatment with antidepressants within 2 weeks prior to the screening,
* had a body mass index greater than 30 kg/m2 and a Child-Pugh score greater than 6 points.
* had made repeated suicide attempts (as assessed by the 12-item Quick Inventory of Depressive Symptomatology scores less than 3),
* had experienced adverse reactions to ketamine or esketamine,
* had known drug use disorders,
* pregnant or breastfeeding

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 435 (Actual)
Dates: Start 2021-02-19 (Actual); Primary Completion 2024-06-23 (Actual); Study Completion 2024-11-27 (Actual)

PRIMARY OUTCOMES:
Depressive symptoms remission | Postoperative 3-day
  Remission is defined as the Montgomery-Åsberg Depression Rating Scale (MADRS) total score no more than 10, MADRS is a sensitive tool used for tracking improvement or progression in patients with major depressive disorder, consisting of 10 items that jointly assess the degree of depressive symptoms.

SECONDARY OUTCOMES:
MADRS scores | Postoperative 3-day
  The differences in MADRS scores
Depressive symptoms response | Postoperative 3-day
  The rates of patients achieving a response
Moderate-to-severe pain | postoperative 3-day
  The rate of severe pain after surgery
Side-effects and Adverse events | During surgery or up to 7 days after surgery
  All drug-related adverse events during surgery or before discharge
Long-term patient outcome | 1, 3, and 6 months after surgery
  The long-term patient outcomes included depressive symptoms and disability as measured by the 12-item World Health Organization Disability Assessment Schedule 2.0 (WHODAS 2.0) at 1, 3, and 6 months after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Ruquan Han, M.D., Ph D., Study Chair — Beijing Tiantan Hospital
Locations (1):
- Beijing Tiantan Hospital, Capital Medical University, Beijing, China

IPD SHARING:
Plan to Share IPD: Yes
The datasets will be available from the primary investigator (Ruquan Han, Email: ruquan.han@ccmu.edu.cn) upon reasonable request after the publication of the study results.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: After the publication of the study results.
Access Criteria: Publication in peer reviewed journal

REFERENCES:
- [Derived] Zhou Y, Ma B, Sun W, Wang J, Fu Y, Wang A, Wang G, Han R. Effect of esketamine on perioperative depressive symptoms in major surgery patients (PASSION II): study protocol for a randomised controlled trial. BMJ Open. 2022 Apr 26;12(4):e056713. doi: 10.1136/bmjopen-2021-056713. PMID 35473735

DOCUMENTS (2):
  • Study Protocol (2021-01-20): https://cdn.clinicaltrials.gov/large-docs/73/NCT04425473/Prot_000.pdf
  • Statistical Analysis Plan (2024-03-15): https://cdn.clinicaltrials.gov/large-docs/73/NCT04425473/SAP_001.pdf